CLINICAL TRIAL: NCT05970458
Title: Stoma Related Complications and Quality of Life Assessment: a Cross-sectional Study With Patients From Ethiopia and Sweden
Brief Title: Stoma Related Complications and Quality of Life Assessments Ethiopia and Sweden
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Åsa Hallqvist Everhov, Principal Investigator, Ass professor, Karolinska Institutet
Other Study IDs: 008/21/Surg
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Stoma Colostomy; Stoma Ileostomy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ethioperm: All patients with a permanent ostomy visiting the stoma center in Addis Abeba
  Interventions: Other: Quality of life assessment
- EthioTemp: All patients waiting for ostomy reversal at Tikur Anbessa Specialized Hospital
  Interventions: Other: Quality of life assessment
- SweSto: All patients visiting the stoma clinic at South General Hospital
  Interventions: Other: Quality of life assessment

INTERVENTIONS:
Other: Quality of life assessment — EQ5D-5L and Stoma QoL

SUMMARY:
Cross-sectional comparative study of general and stoma-specific quality of life in patients with stoma in Addis Abeba, Ethiopia, and Stockholm, Sweden.

DETAILED DESCRIPTION:
Objective: To evaluate the quality of life for patients with ostomy in Ethiopia and Sweden using a general and a specific assessment tool.

Design: Comparative descriptive cross-sectional study. Setting: Tikur Anbessa Specialized Hospital (TASH), Addis Abeba and South General Hospital, Stockholm.

Participants/Exposure: Patients with a permanent ostomy visiting the stoma center in Addis Abeba, patients waiting for ostomy reversal at TASH, and patients visiting the stoma clinic at South General Hospital.

Main outcomes and measure: Quality of life and stoma specific quality of life: EQ5D-5L and Stoma QoL.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥ 18 years old)
* having an ostomy for more than two months
* willingness and ability to give informed consent

Exclusion Criteria:

* non-intestinal stoma

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years old) with ileostomy or colostomy for more than two months, with willingness and ability to give informed consent
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
General quality of life | October 2022 to Jan 2023
  Overall health through visual analogue scale (VAS) from zero (the worst imaginable health) to 100 (the best imaginable health) from the European Quality of Life 5 Dimensions 5 Level Version (EQ5D-5L).
Stoma-specific quality of life | October 2022 to Jan 2023
  The Stoma Quality of life questionnaire consists of 20 questions about stoma-specific aspects of quality of life where each variable is valued equally. Answers are graded in a four-point scale; 1: always, 2: sometimes, 3: rarely, and 4: not at all, with a maximum score of 80. The higher score the better QoL. To get a comparable overall result, the total score (range 20-80) can be converted to a zero to 100 score.

SECONDARY OUTCOMES:
Stoma complications | October 2022 to Jan 2023
  Nipple necrosis, prolapse, parastomal hernia, leakage, itching, bleeding, pain

CONTACTS AND LOCATIONS:
Overall Officials: Åsa Everhov, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Tikur Anbessa Specialized Hospital, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eklov K, Shiferaw A, Rosen A, Bekele S, Ayalew B; ACROSS Collaborative Group; Bringman S, Nygren J, Lofgren J, Everhov AH. Stoma-related complications and quality-of-life assessment: A cross-sectional study with patients from Ethiopia and Sweden. World J Surg. 2024 Jul;48(7):1739-1748. doi: 10.1002/wjs.12209. Epub 2024 May 14. PMID 38743388